CLINICAL TRIAL: NCT01056497
Title: The Effect of A-lipoic Acid (ALA) on Fatty Acid-induced Impairment of Glucose-stimulated Insulin Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Gary Lewis, Professor, Department of Medicine and Physiology, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 090818B; Canadian Diabetes Association
Record Dates: First submitted 2009-12-17; First posted 2010-01-26 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes; Prediabetes
Keywords: diabetes; alpha lipoic acid; endoplasmic reticulum (ER) stress; insulin secretion; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus; Insulin Resistance | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- alpha lipoic acid (Experimental)
  Interventions: Drug: alpha lipoic acid

INTERVENTIONS:
Drug: alpha lipoic acid — A 2 week treatment period with either oral ALA tablets or placebo tablets, followed by 30 hour hospital stay to infuse lipid or saline and to test insulin sensitivity and insulin secretion. For two weeks prior to each admission to hospital and during each hospital admission subjects will ingest 3 tablets 2 times per day with breakfast and supper, 1800mg per day
  Other Names: lipoic acid; ALA

SUMMARY:
Chronically elevated free fatty acids impair insulin sensitivity and insulin secretion (ie lipotoxicity) by a combination of oxidative stress, endoplasmic reticulum (ER) stress and inflammation. This study will test whether alpha-lipoic acid, which has potent antioxidant and anti-inflammatory properties, prevents or ameliorates lipotoxicity.

DETAILED DESCRIPTION:
Alpha-Lipoic Acid (ALA) is a naturally occurring dithiol compound absorbed intact from dietary sources and synthesized enzymatically in the mitochondrion from octanoic acid. It serves a critical role in mitochondrial energy metabolism and is a potent biological antioxidant. It is widely available as an over-the-counter health supplement. It has generated considerable interest among the lay public and the research community for the use of ALA as a nutritive supplement and as a pharmacotherapy for diabetes and many other disorders. There is growing evidence that ALA has beneficial effects on the treatment of type 2 diabetes (T2DM) and some of its complications. It represents an attractive pharmacological target in the treatment of T2DM by modulating the signal transduction pathways in insulin resistance and antagonizing the oxidative and inflammatory stresses, which are major pathways in the pathogenesis of this disorder. Chronic elevation of plasma FFAs are believed to contribute to insulin resistance and defects in insulin secretion by promoting oxidative stress and inflammation. A potent antioxidant and free radical scavenger, ALA also targets cellular signal transduction pathways, which increases glucose uptake and utilization, thus providing specific targeted therapy in the treatment of insulin resistance. ALA has been shown to be safe when taken in high doses (2400mg/d) for prolonged time periods (6 months and longer), even in patients with renal and liver failure. In fact no upper limit for ALA consumption in humans has been established.

* Each subject will undergo 4 studies, 4 to 6 weeks apart. Each study will consist of a 2 week treatment period with either oral ALA tablets or placebo tablets, followed by 30 hour hospital stay to infuse lipid or saline and to test insulin sensitivity and insulin secretion.
* The study will be conducted as a single blind study, with the subject not knowing whether they are receiving a placebo or ALA. For safety reasons and since it will not influence the results of this study it will not be conducted as a double blind study.
* On each of four occasions, 4 weeks apart, after taking the tablets for 2 weeks, the subject will fast overnight for 12-hours prior to their admission to the Toronto General Hospital metabolic research ward for 30 hours to undergo testing as follows. The four studies will be conducted in random order:

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 20-65 years:

1. Written informed consent obtained
2. Body mass index (BMI) > 27kg/m2
3. Glucose tolerance test may be normal or demonstrate impaired glucose tolerance but not frank diabetes
4. Hemoglobin above 130g/L

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL) genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy
3. Type 2 diabetes by history or OGTT
4. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure
5. Any laboratory values: AST > 2x ULN; ALT > 2x ULN; TSH > 6 mU/l
6. A history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions. History of hypersensitivity to heparin
7. Current addiction to alcohol or substances of abuse as determined by the investigator
8. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
9. Any lipid lowering of hypoglycemic agents
10. Previous history of asthma
11. Will not donate blood three months prior to and three months post study procedures
12. Thrombocytopenia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
insulin secretion and insulin sensitivity To determine whether ALA ameliorates or prevents impairment of insulin secretion and insulin sensi | 6 months

SECONDARY OUTCOMES:
To determine the role of oxidative stress and inflammation in the pathogenesis of lipotoxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: gary F Lewis, MD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada